CLINICAL TRIAL: NCT01743469
Title: A Multicentre, Open Label, Early Stopping Design, Proof Of Concept Study With Tasquinimod In Treating Patients With Advanced Or Metastatic Hepatocellular, Ovarian, Renal Cell And Gastric Carcinomas
Brief Title: A Study With Tasquinimod Treating Patients With Hepatocellular, Ovarian, Renal Cell and Gastric Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-55-58102-004; 2012-002326-75 (EudraCT Number)
Record Dates: First submitted 2012-11-29; First posted 2012-12-06 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Advanced or Metastatic Hepatocellular Cancer; Advanced or Metastatic Ovarian Cancer; Metastatic Renal Cell Cancer; Advanced or Metastatic Gastric Carcinoma
Keywords: Advanced; Metastatic; Hepatocellular cancer; Ovarian cancer; Renal cell cancer; Gastric carcinoma
MeSH Terms: conditions — Liver Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell; Stomach Neoplasms; Neoplasm Metastasis | interventions — tasquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hepatocellular Carcinoma Cohort (Experimental): 1 capsule of tasquinimod (0.25 mg or 0.5 mg or 1 mg) taken orally each day until disease progression, lost to follow-up, withdrawal or death.
  Interventions: Drug: Tasquinimod
- Ovarian Carcinoma Cohort (Experimental): 1 capsule of tasquinimod (0.25 mg or 0.5 mg or 1 mg) taken orally each day until disease progression, lost to follow-up, withdrawal or death.
  Interventions: Drug: Tasquinimod
- Renal Cell Carcinoma Cohort (Experimental): 1 capsule of tasquinimod (0.25 mg or 0.5 mg or 1 mg) taken orally each day until disease progression, lost to follow-up, withdrawal or death.
  Interventions: Drug: Tasquinimod
- Gastric Carcinoma Cohort (Experimental): 1 capsule of tasquinimod (0.25 mg or 0.5 mg or 1 mg) taken orally each day until disease progression, lost to follow-up, withdrawal or death.
  Interventions: Drug: Tasquinimod

INTERVENTIONS:
Drug: Tasquinimod — 1 capsule: initially at 0.5 mg/day, increasing to 1 mg/day, maintaining 0.5 mg/day or decreasing to 0.25 mg/day after at least 2 weeks.
  Other Names: ABR-215050
  Arms: Hepatocellular Carcinoma Cohort
Drug: Tasquinimod — 1 capsule: initially at 0.5 mg/day, increasing to 1 mg/day, maintaining 0.5 mg/day or decreasing to 0.25 mg/day after at least 2 weeks.
  Other Names: ABR-215050
  Arms: Ovarian Carcinoma Cohort
Drug: Tasquinimod — 1 capsule: initially at 0.5 mg/day, increasing to 1 mg/day, maintaining 0.5 mg/day or decreasing to 0.25 mg/day after at least 2 weeks.
  Other Names: ABR-215050
  Arms: Renal Cell Carcinoma Cohort
Drug: Tasquinimod — 1 capsule: initially at 0.5 mg/day, increasing to 1 mg/day, maintaining 0.5 mg/day or decreasing to 0.25 mg/day after at least 2 weeks.
  Other Names: ABR-215050
  Arms: Gastric Carcinoma Cohort

SUMMARY:
This was an exploratory proof of concept study to determine the clinical activity of tasquinimod in patients with advanced or metastatic hepatocellular carcinoma, ovarian carcinoma, renal cell carcinoma and gastric carcinoma who had progressed after standard therapies.

DETAILED DESCRIPTION:
This was an early stopping design, Phase II, open label, exploratory proof of concept study to evaluate the activity of tasquinimod in four independent cohorts of patients with different tumour types (patients with hepatocellular, ovarian, renal cell or gastric carcinoma, each with progressive disease after standard therapies). Patients initially received 0.5 mg/day tasquinimod dose, increasing to 1 mg/day after at least 2 weeks, unless there were any individual patient safety and tolerability concerns. The treatment period continued until patient disease progression, lost to follow-up, withdrawal or death. During the treatment period, initial study visits were at Week 2, 4 and 8 (± 2 days) for the hepatocellular carcinoma, the ovarian carcinoma and the renal cell carcinoma cohorts and at Week 2, 4 and 6 (± 2 days) for the gastric carcinoma cohort, to allow careful safety monitoring and to facilitate the identification of the individually tolerated dose. After Week 8, when most patients should have reached their tolerable dose, visit frequency was decreased as follows: at Week 16 and 24 (± 2 days) for the hepatocellular carcinoma, the ovarian carcinoma and the renal cell carcinoma cohorts; and at Week 12, 18 and 24 (± 2 days) for the gastric carcinoma cohort. Thereafter visits were once every 8 weeks (± 2 days) for all cohorts. An end of study treatment/withdrawal (EoST/WD) Visit was to be performed at least 14 days after the last dose of study treatment, and/or before treatment with any alternative antitumour therapy was started. Patients who stopped study treatment before disease progression were to be followed up with tumour imaging every 8 weeks until disease progression. Each patient was subsequently followed up for survival (by visit or telephone call) every 3 months after the EoST/WD Visit until death, lost to follow-up, or withdrawal of consent, or until all surviving patients had been followed-up for at least 9 months after their last administration of study treatment.

The clinical activity of tasquinimod was evaluated independently in each cohort of patients of the four different tumour types. Data were presented as of the following study cut-off dates:

* Hepatocellular carcinoma cohort: 03 December 2014 (efficacy data); 11 April 2016 (safety data).
* Ovarian carcinoma cohort: 27 November 2013 (efficacy data); 05 October 2015 (safety data).
* Renal cell carcinoma cohort: 04 December 2013.
* Gastric carcinoma cohort: 27 September 2013.

ELIGIBILITY:
Inclusion Criteria - All Patients:

1. Able and willing to provide written informed consent and to comply with the study protocol and procedures.
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Life expectancy greater than 3 months in the Investigator's opinion.
5. Disease progression during or after previous cancer treatment.
6. Measurable disease as per Response Evaluation Criteria in Solid Tumours (RECIST) Criteria (v1.1).
7. The following time must have elapsed between previous therapy for cancer and first administration of tasquinimod:

   * At least 2 weeks since previous systemic targeted therapy with small molecule inhibitors, which included any tyrosine-kinase inhibitor.
   * At least 4 weeks since the last dose of systemic anti-cancer therapy other than targeted therapy, which included cytotoxic agents, monoclonal antibody therapy, immunotherapy and prior radiotherapy.
   * At least 1 week since prior hormonal therapy.
   * At least 3 months since prior interferon therapy.
8. Recovery to Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies.
9. At least 4 weeks since any major surgery or open biopsy and 7 days since a core biopsy before first study treatment.
10. Adequate renal function:

    * Creatinine ≤1.5 times upper limit of normal (ULN) or calculated creatinine clearance (CrCl) using the Cockcroft Gault formula ≥60 mL/min, or CrCl ≥60 mL/min.
11. Adequate hepatic function:

    - Serum bilirubin ≤1.5 mg/dL (≤25 μmol/L) for ovarian carcinoma, renal cell carcinoma and gastric carcinoma, serum bilirubin ≤3 mg/dL (≤50 μmol/L) for hepatocellular carcinoma cohorts.
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (≤5 x ULN if liver lesions were present i.e. liver metastasis or primary tumour of the liver for hepatocellular carcinoma cohort).
12. Adequate bone marrow function:

    * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L.
    * Platelets ≥50 x 10^9/L.
    * Haemoglobin ≥90 g/L.
13. Adequate coagulation tests: international normalised ratio (INR) ≤1.5 x ULN.
14. Able to swallow capsules.
15. For women of childbearing potential, a negative pregnancy test must have been documented prior to first administration of study treatment.
16. For women who were not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use adequate methods of contraception (e.g. hormonal implants, combined oral contraceptives, vasectomised partner), during the treatment period and for at least 3 months after the last dose of study treatment.
17. For men: agreement to use a barrier method of contraception during the treatment period and for at least 3 months after the last dose of study treatment.

    Inclusion Criteria - Hepatocellular Carcinoma Cohort:
18. Histologically confirmed and documented hepatocellular carcinoma (excluding fibrolamellar carcinoma).
19. Barcelona Clinic Liver Cancer (BCLC) stage C or BCLC stage B not amenable to locoregional therapy or refractory to locoregional therapy.
20. Liver mass measuring at least 2 cm with characteristic vascularisation seen on either triphasic computed tomography (CT) scan or Magnetic Resonance Imaging (MRI) with gadolinium.
21. At least one measurable or evaluable lesion that was viable (i.e. vascularised), and had not been previously treated with locoregional therapy. A lesion that had been previously treated qualified as a measurable or evaluable lesion if there was demonstrable progression following locoregional therapy.
22. Child-Pugh A Class only.
23. Previously treated with sorafenib. Patients may have experienced radiographically documented disease progression during sorafenib therapy or after discontinuation of sorafenib therapy.
24. The patient had received sorafenib as the most recent systemic therapeutic intervention (any hepatic locoregional therapy that had been administered prior to sorafenib was allowed, but not following sorafenib; radiation to metastatic sites [e.g. bone] following sorafenib therapy was permitted).

Inclusion Criteria - Ovarian Carcinoma Cohort:

18. Histologically confirmed and documented ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer.

19. Progression within 6 months of a platinum containing chemotherapy regimen (i.e. platinum resistant).

20. Progression after up to three lines of chemotherapy.

21. Maximum one line treatment with antiangiogenic therapy.

Inclusion Criteria - Renal Cell Carcinoma Cohort:

18. Metastatic renal cell carcinoma.

19. Histologically or cytologically confirmed and documented renal cell carcinoma with a clear cell component.

20. Previous treatment with at least one vascular endothelial growth factor inhibitor.

21. Disease progression within 6 months prior to first study treatment.

22. Patient had at most two prior targeted therapies for unresectable advanced or metastatic disease.

Inclusion Criteria - Gastric Carcinoma Cohort:

18. Histologically or cytologically confirmed and documented adenocarcinoma of the stomach or gastroesophageal junction.

19. Unresectable advanced or initially metastatic or recurrent after curative resection.

20. Progression after one prior regimen of chemotherapy including fluoropyrimidine and platinum (with or without trastuzumab, if human epidermal growth factor receptor 2 positive [HER2+]).

21. Maximum one line treatment with antiangiogenic therapy.

Exclusion Criteria - All Patients:

1. Other primary malignancy within the past 3 years (except for fully-resected non-melanoma skin cancer, localised prostate cancer with normal prostate specific antigen level, or cervical cancer in situ).
2. Known central nervous system metastasis that was symptomatic and/or required treatment.
3. Malabsorption (other than in patients with gastric carcinoma and partial or complete gastrectomy) or intestinal obstruction.
4. History of pancreatitis.
5. Essential medications that are known potent inhibitors or inducers of CYP3A4.
6. Ongoing treatment with CYP1A2 (including warfarin) or CYP3A4 metabolised drug substance with narrow therapeutic range at the start of study. Treatment with low molecular weight heparin (LMWH) was permitted.
7. History of myocardial infarction, unstable angina, congestive heart failure New York Heart Association class III/IV, cerebrovascular accident, transient ischaemic attack, limb claudication at rest in the previous 6 months, or ongoing symptomatic dysrhythmias, or uncontrolled atrial, or ventricular arrhythmias, or uncontrolled hypertension defined as systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg.
8. Evidence of bleeding diathesis or known coagulopathy.
9. History of venous thromboembolic disease within 3 months prior to first administration of study treatment.
10. The patient had current, severe and uncontrolled medical condition such as infection, diabetes mellitus or other systemic disease.
11. Any condition or illness that, in the opinion of the Investigator or the medical monitor, would have compromised patient safety or interfered with the evaluation of the safety of the drug.
12. Had known positive serology for human immunodeficiency virus.
13. Investigational drug within 28 days or within five times the elimination half-life (whichever was longest) prior to first dose of study treatment.
14. Known allergy to treatment medication or its excipients.
15. Breastfeeding.

Exclusion Criteria - Hepatocellular Carcinoma Cohort:

16. Fibrolamellar carcinoma.

Exclusion Criteria - Ovarian Carcinoma Cohort:

16. Non-epithelial cancer and borderline tumours (e.g. tumours of low malignant potential).

Exclusion Criteria - Gastric Carcinoma Cohort:

16. Other histologic type than adenocarcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (24):
- Belgium (3):
  - Antwerp University Hospital, Wilrijkstraat 10, Edegem
  - Ghent University Hospital, 1K12 IE, De Pintelaan 185, Ghent
  - Leuven cancer institute (LKI), Herestraat, Leuven
- Canada (4):
  - Juravinski Cancer Centre, 699 Concession St, Hamilton, Ontario
  - London Health Sciences Center, 790 Commissoners Road East, London, Ontario
  - Sunnybrook, 2075 Bayview Avenue, Suite T2049, Toronto, Ontario
  - Princess Margaret, 610 University Avenue, Toronto, Ontario
- France (8):
  - Hospital Beaujon, 100 Blvd du Général Leclerc, Clichy
  - Centre Oscar Lambret, 3 rue Frédéric Combemale, Lille
  - Bureau d'Etudes Cliniques du Centre Léon Bérard, 28, rue Laennec, Lyon
  - Hospital Saint-Antoine, 184 rue du Faubourg St Antoine, Paris
  - Hopital Europeen Georges-Pompidou, AP-HP, 20 Rue Leblanc, Paris
  - Centre Eugene Marquis, Avenue bataille Flandres Dunkerque, Rennes
  - Centre René Gauducheau, Boulevard Jacques Monod, Saint-Herblain
  - Institute Gustave-Roussy, 114 rue Edouard Vaillant, Villejuif
- Spain (3):
  - Hospital del mar, Paseo Maritimo 25-29, Barcelona
  - Hospital Gregorio Marañon, Dr. Esquerdo, 44-46, Madrid
  - MD Anderson Cancer Centre, Ctra. Colmenar Viejo Km. 9 100,, Madrid
- United Kingdom (6):
  - Beatson West of Scotland Cancer Centre, 1053 Great Western Road, Glasgow
  - Leicester General Hospital, Gwndolen Road, Leicester
  - The Royal Marsden Hospital, Downs Rd, Sutton, London
  - The Christie Hospital, Wilmslow Road, Withington, Manchester
  - Freeman Hospital, Freeman Road, High Heaton, Newcastle upon Tyne
  - Southampton General Hospital, Tremona Road, Shirley, Southampton

REFERENCES:
- [Derived] Escudier B, Faivre S, Van Cutsem E, Germann N, Pouget JC, Plummer R, Vergote I, Thistlethwaite F, Bjarnason GA, Jones R, Mackay H, Edeline J, Fartoux L, Hirte H, Oza A. A Phase II Multicentre, Open-Label, Proof-of-Concept Study of Tasquinimod in Hepatocellular, Ovarian, Renal Cell, and Gastric Cancers. Target Oncol. 2017 Oct;12(5):655-661. doi: 10.1007/s11523-017-0525-2. PMID 28798986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 24 investigational sites in Belgium, Canada, the United Kingdom, Spain and France. The first patient was enrolled in December 2012 and the study was completed in April 2016.
Pre-assignment Details: In the hepatocellular carcinoma cohort 67 patients were screened, of whom 53 were treated with tasquinimod. In the ovarian carcinoma cohort 63 were screened, of whom 55 were treated. In the renal cell carcinoma cohort 44 were screened, of whom 38 were treated. In the gastric carcinoma cohort 27 were screened, of whom 21 were treated.
Period: Active Treatment Phase
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Started | 53 | 55 | 38 | 21
Completed | 0 | 0 | 0 | 0
Not Completed | 53 | 55 | 38 | 21
Not completed — Adverse Event | 10 | 5 | 8 | 1
Not completed — Disease Progression | 40 | 47 | 30 | 20
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0
Not completed — Missing | 1 | 0 | 0 | 0
Period: Follow-up Period - Post-Treatment
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Started (Entered into follow-up after last treatment with study drug) | 51 | 53 | 37 | 21
Completed | 6 | 5 | 14 | 5
Not Completed | 45 | 48 | 23 | 16
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Death | 43 | 47 | 22 | 16
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All treated patients i.e. all patients who had received at least one dose of tasquinimod.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort | Total
Number analyzed (Participants) | 53 | 55 | 38 | 21 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 34 | 25 | 11 | 89
  >=65 years | 34 | 21 | 13 | 10 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 55 | 10 | 4 | 77
  Male | 45 | 0 | 28 | 17 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 33 | 53 | 33 | 19 | 138
  Unknown or Not Reported | 19 | 2 | 4 | 2 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 0 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 0 | 4
  White | 29 | 49 | 35 | 17 | 130
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 19 | 2 | 3 | 2 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 22 | 9 | 4 | 38
  Belgium | 3 | 10 | 0 | 2 | 15
  United Kingdom | 3 | 11 | 14 | 13 | 41
  France | 43 | 9 | 12 | 2 | 66
  Spain | 1 | 3 | 3 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate, Defined as the Percentage of Patients Who Had Neither Progressed Nor Died as Measured by Centrally Analysed RECIST v1.1 (All Cohorts).
Description: Progression (prog.) defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as a 20% increase in sum of longest diameter of target lesions,or a measurable increase in a nontarget lesion,or appearance of new lesions.
  'Progressed or Died' when time between start of study drug &first date of the following events was ≤ to analysis timepoint +3 days:1) Disease prog. according to central review using RECIST v1.1:date of disease prog. or if missing,first exam date of the visit showing a disease prog.2) Death due to any cause.
  'Neither progressed, nor died' if central assessment by RECIST v1.1 confirmed no disease prog. was observed at the considered timepoint,i.e. time between start of study medication &last examination/visit date of complete response (CR),partial response (PR) or stable disease (SD) ≥ analysis timepoint 7days.In other cases, such as patient withdrawal due to AEs without tumor assessment proving prog.,the patient was considered as 'not assessable'.
Time Frame: Week 12 (Gastric Carcinoma Cohort); Week 16 (Hepatocellular and Renal Cell Carcinoma Cohorts); Week 24 (Ovarian Carcinoma Cohort).
Population: ITT population: All treated patients i.e. all patients who had received at least one dose of tasquinimod. An additional patient was included in the hepatocellular carcinoma cohort, since the 52nd (last patient planned in the protocol) and 53rd were screened at the same time. This 53rd was not included in the primary analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Hepatocellular Carcinoma Cohort; Ovarian Carcinoma Cohort; Renal Cell Carcinoma Cohort; Gastric Carcinoma Cohort: 1 capsule of tasquinimod (0.25 mg or 0.5 mg or 1 mg) taken orally each day until disease progression, lost to follow-up, withdrawal or death.
  1 capsule: initially at 0.5 mg/day, increasing to 1 mg/day, maintaining 0.5 mg/day or decreasing to 0.25 mg/day after at least 2 weeks.
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Number analyzed (Participants) | 52 | 55 | 38 | 21
percentage of participants | 26.9 [15.57 to 41.02] | 7.3 [2.02 to 17.59] | 13.2 [4.41 to 28.09] | 9.5 [1.17 to 30.38]
Statistical Analysis 1: Comparison: Hepatocellular Carcinoma Cohort; The PFS rate was compared with the prespecified threshold (>20%); Test type: Superiority or Other; p = 0.142, Exact binomial test — One-sided alpha of 0.1
Statistical Analysis 2: Comparison: Ovarian Carcinoma Cohort; The PFS rate was compared with the prespecified threshold (>35%); Test type: Superiority or Other; p = 1.000, Exact binomial test — One-sided alpha of 0.1
Statistical Analysis 3: Comparison: Renal Cell Carcinoma Cohort; The PFS rate was compared with the prespecified threshold (>20%); Test type: Superiority or Other; p = 0.800, Exact binomial test — One-sided alpha of 0.1
Statistical Analysis 4: Comparison: Gastric Carcinoma Cohort; The PFS rate was compared with the prespecified threshold (>15%); Test type: Superiority or Other; p = 0.630, Exact binomial test — One-sided alpha of 0.1

2. Secondary Outcome: PFS Rate Measured by Choi Criteria (Hepatocellular Carcinoma Cohort).
Description: PFS rate was defined as the percentage of patients who had neither progressed nor died. Tumour progression was assessed centrally using the Choi criteria.
  Response was measured using the following criteria:
  CR: Disappearance of all lesions, no new lesions; PR: A decrease in size ≥10% or a decrease in tumour attenuation (Hounsfield unit [HU]) ≥15% on CT, no new lesions, no obvious progression of non-measurable disease; SD: Does not meet criteria for CR, PR, or progressive disease (PD), no symptomatic deterioration attributed to tumour progression; PD: An increase in tumour size ≥10% and does not meet criteria of PR by tumour attenuation on CT, new lesions.
Time Frame: Week 16.
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hepatocellular Carcinoma Cohort
Number analyzed (Participants) | 53
percentage of participants | 20.8 [10.84 to 34.11]
Statistical Analysis 1: Comparison: Hepatocellular Carcinoma Cohort; The PFS rate was compared with a prespecified threshold (>20%); Test type: Superiority or Other; p = 0.500, Exact binomial test — One-sided alpha of 0.1

3. Secondary Outcome: Best Overall Response and Response Rates (All Cohorts) Using RECIST v1.1 (Centrally and Locally Analysed).
Description: Best overall response was derived as the best overall response documented before the prespecified timepoint (gastric carcinoma cohort: 12 weeks; Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: Every 6 weeks until Week 24, thereafter, every 8 weeks until disease progression, up to 36 months (gastric carcinoma cohort); every 8 weeks until disease progression, up to 36 months (all other cohorts).
Population: ITT population: all treated patients i.e. all patients who had received at lease one dose of tasquinimod.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Number analyzed (Participants) | 53 | 55 | 38 | 21
percentage of participants
  Best overall response: PR (centrally assessed) | 1.9 [0.05 to 10.07] | 1.8 [0.05 to 9.72] | 0 [NA to NA] — No patients had PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had PR as best overall response, unable to compute 95% CI.
  Best overall response: SD (centrally assessed) | 54.7 [40.45 to 68.44] | 49.1 [35.35 to 62.93] | 47.4 [30.98 to 64.18] | 23.8 [8.22 to 47.17]
  Best overall response: PD (centrally assessed) | 34.0 [21.52 to 48.27] | 41.8 [28.65 to 55.89] | 44.7 [28.62 to 61.70] | 66.7 [43.03 to 85.41]
  Best overall response: NE (centrally assessed) | 9.4 [3.13 to 20.66] | 7.3 [2.02 to 17.59] | 7.9 [1.66 to 21.38] | 9.5 [1.17 to 30.38]
  Response rate (CR or PR) (centrally assessed) | 1.9 [0.05 to 10.07] | 1.8 [0.05 to 9.72] | 0 [NA to NA] — No patients had CR or PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had CR or PR as best overall response, unable to compute 95% CI.
  Best overall response: PR (locally assessed) | 0 [NA to NA] — No patients had PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had PR as best overall response, unable to compute 95% CI.
  Best overall response: SD (locally assessed) | 52.8 [38.64 to 66.70] | 32.7 [20.68 to 46.71] | 39.5 [24.04 to 56.61] | 14.3 [3.05 to 36.34]
  Best overall response: PD (locally assessed) | 43.4 [29.84 to 57.72] | 61.8 [47.73 to 74.59] | 57.9 [40.82 to 73.69] | 81.0 [58.09 to 94.55]
  Best overall response: NE (locally assessed) | 3.8 [0.46 to 12.98] | 5.5 [1.14 to 15.12] | 2.6 [0.07 to 13.81] | 4.8 [0.12 to 23.82]
  Response rate (CR or PR) (locally assessed) | 0 [NA to NA] — No patients had CR or PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had CR or PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had CR or PR as best overall response, unable to compute 95% CI. | 0 [NA to NA] — No patients had CR or PR as best overall response, unable to compute 95% CI.

4. Secondary Outcome: Best Overall Response and Response Rate Based on Choi Criteria (Hepatocellular Carcinoma Cohort).
Description: Per Choi Criteria for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=10% decrease in the sum of the longest diameter of target lesions; Progression, as a 10% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: Every 8 weeks until disease progression, up to 36 months.
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hepatocellular Carcinoma Cohort
Number analyzed (Participants) | 53
percentage of participants
  Best overall response: PR | 20.8 [10.84 to 34.11]
  Best overall response: SD | 32.1 [19.92 to 46.32]
  Best overall response: PD | 34.0 [21.52 to 48.27]
  Best overall response: NE | 13.2 [5.48 to 25.34]
  Response rate (CR or PR) | 20.8 [10.84 to 34.11]

5. Secondary Outcome: Clinical Benefit (All Cohorts).
Description: Clinical benefit was defined as CR, PR or SD lasting at least 12 weeks using centrally or locally assessed RECIST v1.1.
Time Frame: as for outcome 3
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Number analyzed (Participants) | 53 | 55 | 38 | 21
percentage of participants
  Clinical benefit (centrally assessed) | 26.4 [15.26 to 40.33] | 20.0 [10.43 to 32.97] | 15.8 [6.02 to 31.25] | 0.0 [NA to NA] — No patients derived clinical benefit, unable to compute 95% CI.
  Clinical benefit (locally assessed) | 32.1 [19.92 to 46.32] | 16.4 [7.77 to 28.80] | 15.8 [6.02 to 31.25] | 0.0 [NA to NA] — No patients derived clinical benefit, unable to compute 95% CI.

6. Secondary Outcome: PFS From First Study Treatment to Progression or Death Due to Any Cause Based on Choi Criteria (Hepatocellular Carcinoma Cohort).
Description: PFS defined as the time from first study treatment to the first occurrence of a disease progression according to centrally assessed Choi criteria (i.e. increase in tumor size ≥10%) or death due to any cause before initiation of new systemic treatment.
Time Frame: Every 8 weeks until disease progression, up to 36 months.
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hepatocellular Carcinoma Cohort
Number analyzed (Participants) | 53
Weeks | 15.71 [8.00 to 16.43]

7. Secondary Outcome: PFS From First Study Treatment to Progression or Death Due to Any Cause Based on RECIST v1.1 Criteria (All Cohorts).
Description: PFS defined as the time from first study treatment to the first occurrence of a disease progression according to centrally and locally assessed RECIST v1.1 (i.e. increase in tumor size ≥20%) or death due to any cause before initiation of new systemic treatment.
Time Frame: as for outcome 3
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Number analyzed (Participants) | 53 | 55 | 38 | 21
Weeks
  PFS (centrally assessed) | 15.86 [8.00 to 23.14] | 8.00 [7.71 to 17.43] | 14.86 [7.86 to 16.71] | 6.00 [5.29 to 7.29]
  PFS (locally assessed) | 15.71 [8.00 to 16.43] | 7.57 [7.00 to 7.86] | 7.86 [7.29 to 14.71] | 5.79 [5.14 to 6.86]

8. Secondary Outcome: Time to Progression (TTP) by Choi Criteria (Hepatocellular Carcinoma Cohort).
Description: TTP defined as the time from first study treatment to the first occurrence of disease progression defined according to centrally assessed Choi criteria (i.e. increase in tumor size ≥10%) or death due to disease progression before initiation of a new systemic treatment.
Time Frame: Every 8 weeks until disease progression, up to 36 months.
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hepatocellular Carcinoma Cohort
Number analyzed (Participants) | 53
Weeks | 15.86 [8.43 to 16.43]

9. Secondary Outcome: TTP by RECIST v1.1 (All Cohorts).
Description: TTP was defined as the time from first study treatment to the first occurrence of disease progression defined according to centrally and locally assessed RECIST v1.1 criteria (i.e. increase in tumor size ≥20%) or death due to disease progression before initiation of a new systemic treatment.
Time Frame: as for outcome 3
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Number analyzed (Participants) | 53 | 55 | 38 | 21
Weeks
  TTP (centrally assessed) | 15.86 [8.43 to 24.00] | 8.00 [7.71 to 17.43] | 14.86 [7.86 to 16.00] | 6.00 [5.29 to 7.29]
  TTP (locally assessed) | 15.71 [8.00 to 16.43] | 7.57 [7.00 to 7.86] | 7.86 [7.29 to 14.71] | 5.79 [5.14 to 6.86]

10. Secondary Outcome: Overall Survival (OS), Defined as the Time From First Study Treatment to Death Due to Any Cause (All Cohorts).
Description: OS is the time (in weeks) from the first study medication date to death due to any cause. Patients were censored at the date of last contact (the latest between the time of EoST/WD assessment and follow-up visits).
  OS was estimated using Kaplan-Meier analysis.
Time Frame: Time from first study treatment to death, up to 36 months.
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Number analyzed (Participants) | 53 | 55 | 38 | 21
Weeks | 29.29 [25.00 to 38.71] | NA [30.71 to NA] — Median could not be calculated as there was insufficient number of participants with events. | 32.71 [26.43 to 40.86] | 21.57 [13.86 to 33.29]

11. Secondary Outcome: Further Cancer-related Treatment During Follow-up Period (All Cohorts).
Description: Further systemic treatment was coded using World Health Organization (WHO) Drug Dictionary (versions: June 2014 for the hepatocellular carcinoma cohort and June 2013 for the ovarian, renal cell and gastric carcinoma cohorts).
  A frequency table of the number and percentage of patients was provided by Anatomical Therapeutic Chemical (ATC) decode and preferred name.
Time Frame: 16 weeks, Last Patient First Treatment + 16 weeks.
Population: ITT population: all treated patients i.e. all patients who had received at least one dose of tasquinimod.
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
Number analyzed (Participants) | 53 | 55 | 38 | 21
Participants | 16 | 35 | 18 | 8

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected during the active phase of the study from treatment start date until predefined timepoint T2, over approximately 1 year.
Description: Tumour-related signs and symptoms were reported as TEAEs during the study only if they worsened in severity or increased in frequency. Natural progression/deterioration of the malignancy and disease progression that led to death were recorded as part of the efficacy evaluation.
  The Safety population comprised all patients who had received at least one dose of tasquinimod. AEs were coded using MedDRA 17.1 for the Hepatocellular Carcinoma cohort and version 16.1 for all other cohorts.
Arm/Group | Hepatocellular Carcinoma Cohort | Ovarian Carcinoma Cohort | Renal Cell Carcinoma Cohort | Gastric Carcinoma Cohort
All-Cause Mortality (participants affected / at risk) | 38/53 | 22/55 | 22/38 | 16/21
Serious Adverse Events (participants affected / at risk) | 14/53 | 19/55 | 11/38 | 7/21
Other Adverse Events (participants affected / at risk) | 53/53 | 55/55 | 38/38 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatocellular Carcinoma Cohort (N=53) | Ovarian Carcinoma Cohort (N=55) | Renal Cell Carcinoma Cohort (N=38) | Gastric Carcinoma Cohort (N=21)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammatory myofibroblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatocellular Carcinoma Cohort (N=53) | Ovarian Carcinoma Cohort (N=55) | Renal Cell Carcinoma Cohort (N=38) | Gastric Carcinoma Cohort (N=21)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (2)
Oedema peripheral (General disorders) | 16 (18) | 17 (21) | 4 (9) | 2 (2)
Fatigue (General disorders) | 31 (36) | 31 (41) | 7 (7) | 15 (18)
Asthenia (General disorders) | 7 (8) | 5 (7) | 11 (17) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 8 (10) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (11) | 9 (10) | 6 (6) | 6 (6)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0) | 3 (4)
Weight decreased (Investigations) | 13 (14) | 3 (3) | 5 (5) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (3) | 6 (7) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 6 (7) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 9 (9) | 3 (3) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 12 (12) | 9 (10) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 12 (13) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 10 (13) | 4 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 4 (5) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 15 (17) | 19 (20) | 8 (8) | 9 (11)
Nausea (Gastrointestinal disorders) | 21 (28) | 24 (30) | 12 (13) | 13 (17)
Vomiting (Gastrointestinal disorders) | 18 (25) | 16 (21) | 9 (9) | 13 (18)
Constipation (Gastrointestinal disorders) | 15 (16) | 12 (12) | 13 (13) | 11 (13)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (6) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 14 (20) | 14 (18) | 7 (8) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 10 (12) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 13 (14) | 1 (1) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Ascites (Gastrointestinal disorders) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 3 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 14 (15) | 5 (6) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (6) | 4 (6) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 10 (11) | 2 (3) | 3 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5) | 4 (6) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (6) | 4 (4) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 21 (22) | 20 (25) | 11 (11) | 15 (17)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 6 (6) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 7 (7) | 0 (0) | 2 (3)
Rash pustular (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor required reasonable opportunity to review any abstract, presentation, or paper before the material was submitted for publication or communicated. This also applied to any amendments that were requested by referees or journal editors. The Sponsor committed to comment on the draft documents within a time period agreed in the contractual arrangements between the Sponsor and authors or their institution. Delays were also possible if publication would adversely affect patentability.